CLINICAL TRIAL: NCT01471821
Title: Study to Evaluate the Activity and Tolerability of Lopinavir/Ritonavir and Lamivudine Bitherapy Instead of a Triple Therapy That Includes Lopinavir/Ritonavir and Lamivudine or Emtricitabine in HIV Patients With Viral Suppression: Controlled Clinical Trial, Open Label, Randomized, of 48 Weeks of Follow-up
Brief Title: Study to Evaluate the Activity and Tolerability of Lopinavir/Ritonavir and Lamivudine Bitherapy in HIV Patients With Viral Suppression
Acronym: OLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, Clinical Trial Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OLE
Record Dates: First submitted 2011-11-15; First posted 2011-11-16 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- simplification (Experimental): Lopinavir/ritonavir (400/100 BID) plus lamivudine (300 QD)
  Interventions: Drug: antiretroviral treatment
- Continue with current treatment (Active Comparator)
  Interventions: Drug: antiretroviral treatment

INTERVENTIONS:
Drug: antiretroviral treatment — antiretroviral treatment

SUMMARY:
This is a prospective, open controlled trial in which HIV-1 with viral suppression patients will be randomized to continue with their current treatment (lopinavir/ritonavir plus emtricitabine or lamivudine plus any nucleoside analogue reverse transcriptase inhibitor) or to simplify to lopinavir/ritonavir plus lamivudine.

Randomization will be stratified according to the values of nadir CD4 and time of viral suppression.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex (female or male) and 18 years or older.
* Patients seropositive for HIV-1 using standard diagnostic criteria.
* There is confirmation of viral load to be lower than 50 cop/ml during the 6 previous months to inclusion. The requirement is to have at least two viral loads lower than 50 cop/mL separated by 6 months and no one >50cop/mL during the 6 months before inclusion.
* Patients on continuous HAART consisting of LPV/r, emtricitabine (FTC) or 3TC (lamivudine) and an NRTI for at least 2 months before being randomized in this study.
* Patients who are clinically stable, in the opinion of the investigator, at entry into the study (clinical status and chronic medication must not have not been modified at least 14 days prior to randomization). Patients receiving therapy for an active opportunistic infection are eligible for enrollment if the above criteria are met. Standard prophylaxis of opportunistic infections is permitted.

Exclusion Criteria:

* Pregnancy, nursing, or planned pregnancy during the study period.
* Previous failure with regimens including a protease inhibitor (PI) or 3TC/FTC.
* Known resistance mutations to PIs or 3TC/FTC.
* Patients with an active opportunistic infection or malignancy. Patients with a stable chronic opportunistic infection may be included in the study.
* Any disease or history of disease which, in the opinion of the investigator, might confound the results of the study or pose additional risk to patient treatment.
* Patients diagnosed with visceral Kaposi's sarcoma (KS), patients with lymphoedema secondary to cutaneous KS or cutaneous or palatine KS who have been treated with systemic immunosuppressive therapy must also be excluded.
* Patients with chronic hepatitis B on treatment with tenofovir + 3TC/FTC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with no treatment failure | 48 weeks
  * viral failure, defined as two viral loads above 50 copies/ml at least two weeks apart
  * death
  * developing new CDC-C events
  * withdrawing consent
  * being lost to follow-up
  * switching assigned treatment for any cause

SECONDARY OUTCOMES:
Proportion of patients with no viral failure | 48 weeks
  defined as two viral loads above 50 copies/ml. Patients lost to follow-up or changing treatment will not be taken into account for this analysis
Proportion of patients with no therapeutical failure | 48 weeks
  defined as in the primary outcome but with two viral loads above 400 copies/ml, not 50 as in the primary outcome.
Proportion of patients with no viral failure | 48 weeks
  defined as two viral loads above 400 copies/ml
Time to viral failure | 48 weeks
  Two different analysis will be carried out: with 50 copies/ml threshold and with 400 copies/ml threshold
Proportion of patients with blips | 48 weeks
  Defined as one viral load above 50 and below 400 copies/ml with next viral load below 50 copies/ml
Change from baseline CD4 | 48 weeks
Lipidic profile change from baseline | 48 weeks
Creatinine clearance change from baseline | 48 weeks
Proportion of patients with proximal tubular renal disfunction | 48 weeks
Lipodystrophy changes from baseline | 48 weeks
  evaluated using two questionnaires: lipoatrophy and fat accumulation
Adherence to treatment | 48 weeks
Mortality and progression to AIDS | 48 weeks
Adverse events per treatment branch | 48 weeks
Proportion of patients switching study treatment due to an adverse event | 48 weeks
Proportion of serious adverse events related to treatment | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: José Ramón Arribas, MD, Principal Investigator — Hospital Uniuversitario La Paz
Locations (2):
- Spain (2):
  - Hospital Clínic i Provincial Barcelona, Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid, Madrid

REFERENCES:
- [Derived] Arribas JR, Girard PM, Landman R, Pich J, Mallolas J, Martinez-Rebollar M, Zamora FX, Estrada V, Crespo M, Podzamczer D, Portilla J, Dronda F, Iribarren JA, Domingo P, Pulido F, Montero M, Knobel H, Cabie A, Weiss L, Gatell JM; OLE/RIS-EST13 Study Group. Dual treatment with lopinavir-ritonavir plus lamivudine versus triple treatment with lopinavir-ritonavir plus lamivudine or emtricitabine and a second nucleos(t)ide reverse transcriptase inhibitor for maintenance of HIV-1 viral suppression (OLE): a randomised, open-label, non-inferiority trial. Lancet Infect Dis. 2015 Jul;15(7):785-92. doi: 10.1016/S1473-3099(15)00096-1. Epub 2015 Jun 7. Erratum In: Lancet Infect Dis. 2015 Aug;15(8):875. doi: 10.1016/S1473-3099(15)00112-7. PMID 26062880